CLINICAL TRIAL: NCT01913691
Title: Phase II Open-Label Trial of Ipilimumab for Metastatic Merkel Cell Carcinoma
Brief Title: Study of the Drug Ipilimumab for Metastatic Merkel Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130173; 13-C-0173
Record Dates: First submitted 2013-07-28; First posted 2013-08-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-03

CONDITIONS: Merkel Cell Carcinoma
Keywords: Neuroendocrine Skin Cancer; Merkel Cell Polyomavirus; Immunotherapy
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab is a recombinant, human monoclonal antibody that binds to CTLA-4. It is commercially available under the brand name Yervoy . The use of ipilimumab for MCC is investigational: a study-specific supply of medication will be provided by Bristol-Myers Squibb.

SUMMARY:
Background:

- Ipilimumab is a drug used to treat melanoma that cannot be treated surgically. It targets a molecule found on T-cells in the human immune system. Blocking these molecules on the T-cells might allow the cells to help destroy melanoma cells more effectively. This drug has also been studied in other cancers such as prostate cancer and lung cancer, but not yet in Merkel cell carcinoma (MCC). Researchers think therapy like ipilimumab that enhances the immune system may be effective against MCC. They want to study how safe the drug is and its effect on the immune system and tumors.

Objectives:

- To determine the number of subjects with MCC who take the study drug that remain alive 12 months later.

Eligibility:

- Adults 18 years and older who have metastatic MCC.

Design:

* Participants will be screened with a medical history and physical exam.
* Participants will receive the study drug 4 times, one dose every 21 days. After the 4 visits, participants will receive a maintenance dose of the drug every 12 weeks until the drug is no longer beneficial.
* They will receive the drug through a plastic tube usually inserted in a vein on the arm.
* It will take 90 minutes to give each dose.
* At all visits, participants will be screened with a medical history, physical exam, and blood tests. Any tumors on their skin will be measured and photographed.
* Every 12 weeks during the study and maintenance period, participants will have a CT scan. Throughout the study and maintenance period, they will have blood and skin tests.

DETAILED DESCRIPTION:
Background:

Merkel cell carcinoma (MCC) is a rare, aggressive neuroendocrine cancer of the skin with a mortality of approximately 33%. Approximately one-third of patients present with metastatic disease, for which there is no effective treatment. Merkel cell polyomavirus (MCV), a DNA virus that expresses T antigen oncoproteins, was found to be clonally integrated into the genome of the majority of MCC tumors. MCC tumor progression is believed to be associated with the development of immune evasion, and multiple lines of evidence (higher incidence in immunocompromised populations, reports of spontaneous regression, responses to immune modulators, and improved prognosis associated with CD8+ intratumoral lymphocytes) suggest that immunotherapy may improve outcomes in patients with advanced MCC. Ipilimumab is a recombinant, human monoclonal antibody that binds to cytotoxic Tlymphocyte- associated antigen 4 and has shown efficacy in metastatic melanoma.

Objectives:

Primary:

-Determine overall survival at 12 months.

Secondary:

* Determine the best overall response rate, as assessed by modified RECIST immunerelated response criteria, at week 12.
* Determine median survival.
* Determine disease-specific survival (DSS) and progression-free survival (PFS).
* Evaluate the safety and tolerability of ipilimumab in patients with metastatic MCC.
* Assess biomarkers of immune activation and MCV-specific immune response.

Eligibility:

* Patients (age greater than or equal to 18 years) with metastatic MCC (AJCC stage 3b or 4).
* Immunocompromised individuals and patients with autoimmune disease are excluded.

Design:

* Patients will enroll at the NIH Clinical Center, Bethesda, MD (primary site) or at a study sub-sites Memorial Sloan-Kettering Cancer Center, New York, NY; University of Michigan, Ann Arbor, MI; or University of Pennsylvania, Philadelphia, PA.
* Ipilimumab will be given at a dose of 10 mg/kg as a 90-minute intravenous infusion on day 1 of each 21-day cycle for 4 cycles. After 4 doses, patients may receive a maintenance dose every 12 weeks until disease progression or unacceptable toxicity, for up to an additional 4 doses.
* Imaging scans will be done at week 12, and every 12 weeks on study starting week 21.
* Patients will remain on-study for follow-up for 96 weeks after the last of the initial 4 doses.
* Response and progression will be evaluated using modified RECIST immune-related response criteria.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of Merkel cell carcinoma confirmed by the Laboratory of Pathology, NCI, or the participating institute s Department of Pathology.
* Unresectable or metastatic Merkel cell carcinoma
* Measurable disease as defined by lesions that are measured in at least one dimension >20mm by CXR, as > 10mm with CT scans, or > 10mm with calibers by clinical exam.
* Life expectancy greater than or equal to 6 months.
* ECOG performance status of 0-2
* Willing to travel to the NIH or study sub-sites (MSKCC, UMich, or Penn) for follow-up visits.
* Patients must have recovered from acute toxicities related to prior therapy or surgery.
* Patients must receive at least one line of chemotherapy and achieve partial response(30% reduction in tumor burden) or better prior to enrollment. EXCEPTION: Patients with asymptomatic tumors showing no or minimal progression (<20% tumor burden) within the last 2 months can be enrolled without prior chemotherapy.
* Age greater than equal 18 years. Because no dosing or adverse event data are currently available on the use of ipilimumab in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Patients must have adequate hematological, hepatic, and renal laboratory values, as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL

    -----total bilirubin within normal institutional limits (except subjects with Gilbert s Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
  * AST(SGOT)/ALT(SGPT) <2.5 times institutional upper limit of normal
  * creatinine <2.0 times institutional upper limit of normal.
* The effects of ipilimumab on the developing human fetus are unknown. For this reason and because ipilimumab was found to have teratogenic and abortifacient effects in animal studies, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after the last injection of ipilimumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Prior treatment with ipilimumab.

-Patients who are immunocompromised as listed:

* Human immunodeficiency virus infection, or Hepatitis B or C infection, due to the unknown effects of ipilimumab on viral replication and immune function and the potential for severe side effects.
* Chronic administration (defined as daily or every other day for continued use >14 days) of systemic corticosteroids (including steroid eye drops) or other immune suppressive drugs, within 14 days of the first planned dose of ipilimumab. Nasal, or inhaled steroid, and topical steroid creams for small body areas are not excluded.
* Patients who have undergone allogeneic peripheral stem cell transplantation, or solid organ transplantation requiring immunosuppression

Prior Splenectomy

-Patients with history of, or active autoimmune disease that has required treatment, such as Addison's disease, autoimmune thyroiditis, Grave s disease, systemic lupus erythematous, rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barr(SqrRoot)(Copyright) syndrome), Goodpasture syndrome, ulcerative or hemorrhagic colitis, autoimmune hypophysitis/hypopituitarism, and autoimmune hemolytic anemia.

EXCEPTIONS: Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including CNS, heart, lungs, kidneys, skin, and GI tract will not be excluded. Patients with type 1 diabetes mellitus, or vitiligo, or endocrine deficiencies such as hypothyroidism will not be excluded if the condition is well controlled.

* Other active malignancies within the past 12 months. EXCEPTIONS: Patients with adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix or bladder will not be excluded. Patients with low or intermediate-risk CLL (Rai stage 0-II, Binet stage A or B) without progressive or symptomatic disease, who are being monitored without therapy will not be excluded.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke < 6 months prior to enrollment, myocardial infarction < 6 months prior to enrollment, unstable angina, or congestive heart failure ( (Bullet) NYHA III).
* Pulmonary disease which, in the opinion of the investigator, may impair the patient's respiratory tolerance to the study drug (e.g., interstitial lung disease, severe chronic obstructive pulmonary disease).
* Presence of serious or life-threatening intercurrent medical illness.
* Patients with symptomatic or progressive (progression within the last 3 months) brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Pregnant women are excluded from this study because, based on animal studies, ipilimumab has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ipilimumab, breastfeeding should be discontinued if the mother is treated with ipilimumab.
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints.
* Receipt of chemotherapy or an investigational agent within 21 days (or 60 days for an antibody-based therapy) of the first planned dose of study drugs.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-09; Primary Completion 2014-02-03 (Actual); Study Completion 2014-02-03 (Actual)

PRIMARY OUTCOMES:
Overall survival at 12 months with ipilimumab treatment. | 1 year

SECONDARY OUTCOMES:
Determine the best overall response rate, median survival, disease-specific survival, and progression free survival. | 12 weeks
Determine median survival, disease-specific survival, and progressionfree survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Isaac F Brownell, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Hodgson NC. Merkel cell carcinoma: changing incidence trends. J Surg Oncol. 2005 Jan 1;89(1):1-4. doi: 10.1002/jso.20167. PMID 15611998
- [Background] Agelli M, Clegg LX. Epidemiology of primary Merkel cell carcinoma in the United States. J Am Acad Dermatol. 2003 Nov;49(5):832-41. doi: 10.1016/s0190-9622(03)02108-x. PMID 14576661
- [Background] Lemos B, Nghiem P. Merkel cell carcinoma: more deaths but still no pathway to blame. J Invest Dermatol. 2007 Sep;127(9):2100-3. doi: 10.1038/sj.jid.5700925. PMID 17700621